CLINICAL TRIAL: NCT05058170
Title: Characterization of Renal Allograft Fibrosis and Prediction of Outcome Using a Quantitative MRI Approach
Brief Title: Renal Allograft Fibrosis Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Weill Medical College of Cornell University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sara Lewis, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 20-2690; R01DK129888 (NIH)
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Renal Allograft Fibrosis
Keywords: Renal allograft fibrosis; Kidney; Chronic Kidney Disease; Transplant; MRI
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples will be collected at both centers for standard of care urinalysis and mRNA biomarker profiling.
  Urine samples with mRNA Urine will be collected to measure CD3 mRNA, CXCL10 mRNA, CDH1 mRNA, SLC12A1 mRNA, and Vim mRNA and other urine biomarkers. The research team will not perform whole genome sequencing as part of this study.
  Blood will be collected for GFR
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Renal transplant patients

SUMMARY:
Despite the reduction in acute rejection episodes in renal transplant patients due to modern immunosuppression, proportionate improvements in long-term allograft survival have not been achieved. Virtually any disease or injury affecting renal allografts can culminate in irreversible injury of tubular epithelial cells and the development of interstitial fibrosis and tubular atrophy (IFTA). Renal allograft fibrosis drives chronic kidney disease (CKD) progression, predicts allograft failure and is associated with increased patient mortality. Other prognostic and/or actionable diagnoses described by the pathologic Banff scheme, such as inflammation, often co-exist and contribute to IFTA. Immune cell infiltration within allografts and within areas of IFTA (i-IFTA) can drive progressive kidney injury, fibrosis and worsened outcome. Pathology is the reference standard for IFTA; however, allograft biopsy has many well-known limitations and is not an ideal method for monitoring patients during trials of new therapies aimed at improving allograft survival. There is an urgent and unmet need for non-invasive assessment of renal allograft IFTA.

Multiparametric MRI (mpMRI), including relaxometry [the spin-lock relaxation time T1ρ, a marker of interaction of water with macromolecules in tissues; the spin-lattice relaxation time T1, a marker of interstitial edema and collagen volume fraction)] and advanced diffusion [intravoxel incoherent motion diffusion-weighted imaging (IVIM-DWI), a marker of diffusion and perfusion] provides insight into renal structure and function. Validation of advanced MRI methods as markers of renal allograft IFTA would be of major clinical significance to enable early detection, assess the efficacy of novel anti-fibrotic agents, and provide longitudinal disease monitoring. The study team has established proof-of-concept in renal allografts with stable function and IFTA without confounding rejection or infection that mpMRI techniques are feasible for measuring fibrosis, especially using the combination of T1 and DWI. The study has established that urinary biomarkers for renal allograft fibrosis are also promising and have been validated against pathology in initial studies.

In this proposal, the researchers will develop a short, non-contrast multiparametric MRI (mpMRI) protocol, consisting of advanced relaxometry (T1 mapping and T1ρ) and advanced diffusion weighted imaging (IVIM-DWI) to accurately detect and stage allograft fibrosis, taking into account confounding Banff variables of inflammation and tested against biopsy. The researchers will also assess the added value of urinary biomarkers of IFTA and if successful, this study will benefit a large population of patients with renal allograft fibrosis in the United States, enabling early diagnosis, optimized treatment planning, prognostication and longitudinal disease monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients post renal transplantation, with acute or chronic allograft dysfunction, referred for biopsy based on clinical grounds (indication biopsy). Patients with be considered to have allograft dysfunction if: 1. Patients will be considered to have acute allograft dysfunction if there is a 15% decline in eGFR or a 0.3-mg/dL increase in sCr level, with laboratory and clinical findings that exclude pre-renal or post-renal dysfunction. 2. Patients will be considered to have chronic allograft dysfunction if there is a sustained >50% increase in sCr/decrease in eGFR (over their post-transplant nadir creatinine), occurring over a period of >3 months, with laboratory and clinical findings that exclude pre-renal or post-renal dysfunction.
* Patients with stable allograft function and donor-specific antibody (DSA) positivity, referred for surveillance biopsy at 3 and 12 months post transplantation. Patients with be considered to have stable allograft function if: 1. Patients will be considered to have chronic stable allograft function if they have a stable eGFR > 45 ml/min & a spot urine protein:creatinine ratio < 0.2; 2. Stable creatinine/eGFR (i.e. <25% change in serum creatinine (Cr) and/or eGFR from post transplant baseline).
* Patient is able to give informed consent for this study.
* Study team will recruit patients after 1 month post-transplant period since the early post transplant course is associated with increased risk of acute dysfunction (i.e. acute tubular necrosis or acute rejection episodes).
* Healthy volunteers with no renal disease will be recruited for protocol optimization and to serve as controls.
* Potential renal donors undergoing clinical non-contrast or contrast-enhanced MRI will be recruited to serve as controls.

Exclusion Criteria:

* Age less than 18 years.
* Renal transplantation <1 month prior to scanning.
* Evidence of large vessel or urinary tract complication of the renal transplant.
* Unable or unwilling to give informed consent.
* Contra-indications to MRI

  1. Electrical implants such as cardiac pacemakers or perfusion pumps.
  2. Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants.
  3. Ferromagnetic objects such as jewelry or metal clips in clothing.
  4. Pregnant subjects.
  5. Pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions.

The inclusion and exclusion criteria are identical at ISMMS and WCMC.

* Screening for eligibility will be performed by the transplant nephrology team at both centers. Data relevant to eligibility will be reviewed, including age, presence of allograft dysfunction and its ascertainment (clinical, laboratory and prior biopsy data), and MRI safety will also be reviewed by the study coordinator.
* There are no exclusions based on race, sex/gender, preferred language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed renal allograft fibrosis.
Sampling Method: Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Presence of renal allograft fibrosis | 2 weeks after renal allograft biopsy
  Detection of the presence of renal allograft fibrosis using MRI in patients undergoing biopsies.
Banff scoring system for fibrosis | 2 weeks after renal allograft biopsy
  Detection of the severity of renal allograft fibrosis using MRI in patients undergoing biopsies, using the Banff scoring system for interstitial fibrosis (ci) + tubular atrophy (ct); each subscore from 0-3 with full range from 0-6, higher score indicates higher severity).

SECONDARY OUTCOMES:
Presence of renal allograft inflammation | 2 weeks after renal allograft biopsy
  Detection of the presence of renal allograft inflammation using MRI in patients undergoing biopsies.
Banff scoring system for inflammation | 2 weeks after renal allograft biopsy
  Detection of the severity of renal allograft inflammation using MRI in patients undergoing biopsies using the Banff scoring system. the Banff lesion scored include inflammation in the area of IFTA (i-IFTA), tubulitis (t), glomerular basement membrane (GBM) double contours (cg), vascular fibrous intimal thickening (cv), glomerulitis (g), intimal arteritis (v), and peritubular capillaritis (ptc), all subscores range, 0-3, with full range 0-3, higher score indicating higher severity.
4-gene fibrosis signature score | Within 1 year of urine processing
  4-gene fibrosis signature score as a measurement of urinary mRNA (which consists of CDH1 mRNA, SLC12A1 mRNA, Vim mRNA and 18S rRNA) obtained from urine cells for the detection of renal allograft fibrosis. Measurement is a continuous scale with no maximum, higher score indicates higher severity.
3-gene inflammation score | Within 1 year of urine processing
  3-gene inflammation score as a measurement of urinary mRNA (which consists of CD3 mRNA, CXCL10 mRNA, and 18S rRNA) obtained from urine cells for the detection of renal allograft inflammation. Measurement is a continuous scale with no maximum, higher score indicates higher severity.
Change in estimated Glomerular filtration rate (eGFR) | Baseline and within 2 years after initial MRI
  Renal function assessed by estimated Glomerular filtration rate (eGFR) which is a test used to check how well the kidneys are working. Specifically, it estimates how much blood passes through the glomeruli each minute. Glomeruli are the tiny filters in the kidneys that filter waste from the blood.
Change in Protein level in urine | Baseline and within 2 years after initial MRI
  Renal function assessed by protein level in urine to detect proteinuria. Proteinuria is defined as (>1 g/dL).
Change in Interstitial fibrosis and tubular atrophy (IFTA) stage | Within 2 years after initial MRI
  Renal function assessed by change in IFTA stage as determined by the Banff scoring system. The Banff lesion score include interstitial fibrosis (ci) + tubular atrophy (ct). Each subscore range 0-3, with total range from 0-6 and a higher score indicates higher severity.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lewis, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Octavia Bane, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Weill Cornell Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No
Not encompassed in the grant proposal to share data with others outside of this study.